CLINICAL TRIAL: NCT03286530
Title: Phase II Study of Maintenance Ruxolitinib After Allogeneic Stem Cell Transplantation for Older Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) in Complete Remission
Brief Title: Ruxolitinib + Allogeneic Stem Cell Transplantation in AML
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Washington University School of Medicine (Other); Vanderbilt University (Other); Ohio State University (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Gabriela Hobbs, Prinicipal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-273
Record Dates: First submitted 2017-08-09; First posted 2017-09-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia in Remission; Allogeneic Stem Cell Transplantation
Keywords: Acute Myeloid Leukemia; Acute Myeloid Leukemia in Remission; Allogenic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Following a standard of care allogeneic stem cell transplantation, participants will be started on Ruxolitinib. Ruxolitinib is administered orally 2 times per day at a fixed dose. Each study treatment cycle lasts 28 days. Up to 24 cycles.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Patients who fulfill eligibility criteria will be entered into the trial to receive Ruxolitinib.
  After the screening procedures confirm participation in the research study. The participant will be given a drug diary. The participant will be asked to document information in the drug diary about the study treatment.
  Other Names: Jakafi

SUMMARY:
This research study is studying a drug that may help decrease the chances of relapse after Allogeneic Stem Cell transplantation for Acute Myeloid Leukemia. The name of the study drug involved in this study is:

• Ruxolitinib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ruxolitinib for this specific disease but it has been approved for other blood diseases.

In this research study, investigators are trying to discover if ruxolitinib will decrease chances of relapse after having an allogeneic stem cell transplantation.

Ruxolitinib is a medication that blocks certain proteins called tyrosine kinases. Specifically, it blocks tyrosine kinases called JAK2. Many cancers have over active "cell signaling." What this means is that certain functions in the cancer cells never turn off and this makes them grow in an uncontrolled way. Ruxolitinib, shuts down the pathway that depends on the JAK2 tyrosine kinases. The JAK2 pathway is over active with acute myeloid leukemia. Ruxolitinib has also been shown to lower the rates of graft versus host disease, a complication of transplant. The exact way ruxolitinib does this is not yet clear but it may have to do with its ability to block the JAK2 pathway since this pathway can also lead to inflammation in the body.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have pathologically confirmed AML in CR1 as defined by:

  * Bone marrow biopsy with < 5% blasts
  * No clusters or collections of blast cells
  * No extramedullary leukemia
  * Absolute neutrophil count ≥ 1000/µL (achieved post-induction at some point)
  * Please note that full platelet recovery is not necessary, and thus, patients achieving CRp are eligible.

    ---Or participants have pathologically confirmed MDS as defined by:
  * Bone marrow biopsy with <10% blasts
  * Patients receiving MDS-directed therapy must be off treatment for > 2 weeks prior to start of conditioning.
* Participants must be designated to undergo reduced intensity allogeneic peripheral blood hematopoietic stem cell transplantation (HCT). Consent will be obtained prior to admission for HCT. The following HCT conditions must be planned:

  * Donors must be 8/8 HLA-matched (at the allele level) as defined by matching at HLA-A, -B, -DR and -C who pass institutional standard to serve as a peripheral blood stem cell donor
  * Donor grafts must be G-CSF mobilized peripheral blood stem cells with dose and apheresis logistics at the discretion of institutional standard
  * Conditioning therapy will be one of the following 3 options:

    * Fludarabine / Melphalan where fludarabine is ≥ 90 mg/m2 IV total dose and melphalan is 100-140 mg/m2 IV total dose. Exact logistics of administration are at the discretion of institutional standard.
    * Fludarabine / Busulfan where fludarabine is ≥ 90 mg/m2 IV total dose and busulfan = 6.4 mg/kg IV total dose. Exact logistics of administration are at the discretion of institutional standard.
    * Fludarabine / Busulfan where fludarabine is ≥ 90 mg/m2 IV total dose and busulfan is dosed to achieve AUC of 4000 µmol/min based on a pharmacokinetics determined from a test dose. Exact logistics are at the discretion of institutional standard.
    * GVHD prophylaxis is comprised of tacrolimus / short course methotrexate as defined by tacrolimus started prior to day 0 of HCT and methotrexate given after HCT on days +1, +3 and +6 ± +11 at a dose of 5-10 mg/m2 IV. Exact logistics are at the discretion of the treating institution.
* Age ≥ 60 and ≤ 80 years old
* ECOG performance status 0-2
* Male participants must agree to use an acceptable method for contraception during the entire study treatment period and through 6 months after the last dose of treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have had a prior allogeneic HSCT.
* Patients without normal organ function defined as follows:

  * AST (SGOT), ALT (SGPT) and Alkaline Phosphatase >3 × institutional Upper Limit of Normal (ULN)
  * Direct bilirubin >2.0 mg/dL
  * Adequate renal function as defined by calculated creatinine clearance ≤ 40 mL/min (Cockcroft-Gault formula)
* Have a history of other malignancy(ies) unless:

  * They have been disease-free for at least 5 years and are deemed by the treating investigator to be at low risk for recurrence of that malignancy,

    --- or
  * The only cancer they have had is cervical cancer in situ, or basal cell or squamous cell carcinoma of the skin
* Have a chronic or active infection that requires systemic antibiotics, antifungal or antiviral treatment.
* Have current or a history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 40%, as measured by MUGA scan or echocardiogram)
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Be HIV-positive
* Have a systemic infection requiring IV antibiotic therapy, nor any other severe infection
* Planned use of ex vivo or in vivo T-cell depletion
* Have current or a history of ventricular or life-threatening arrhythmias or diagnosis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1-year GVHD/relapse free survival rate (GRFS rate) | 1 Year
  The number of participants surviving after one year that have not experienced graft-versus-host disease (GVHD) or graft relapse (GRFS rate).

SECONDARY OUTCOMES:
Progression Free Survival | Until disease progression or death from any cause, approximately 5 years
  Kaplan-Meier estimates of progression free survival (PFS) will be calculated, with patients without an event being censored at last date of contact
Overall Survival | Until death, approximately 5 years
  Overall survival is measured as the time from the hematopoietic stem cell transplantation (HSCT) until death. Participants without an event will be censored at the date of last contact.
Cumulative incidence of drug related toxicities | 2 Years
  Cumulative incidence of treatment related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE 4). Early deaths from all other causes are considered a competing risk.
Time to Relapse | 2 Years
  The amount of time from the hematopoietic stem cell transplantation (HSCT) until disease relapse. Relapse is the recurrence of cancer after having a bone marrow biopsy without evidence of cancer. Time to treatment-related mortality is considered a competing risk.
Time to treatment-related mortality (TRM) | 2 Years
  The amount of time between receiving the HSCT and death due to a treatment related cause. Time to relapse is considered a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriell Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Medical College of Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeFilipp Z, Kim HT, Knight LW, O'Connor SM, Dhaver SE, White M, Dholaria B, Schroeder MA, Vasu S, Abedin S, Chung J, El-Jawahri A, Frigault MJ, McAfee S, Newcomb RA, O'Donnell PV, Spitzer TR, Chen YB, Hobbs GS. Low rates of chronic graft-versus-host disease with ruxolitinib maintenance following allogeneic HCT. Blood. 2025 May 15;145(20):2312-2316. doi: 10.1182/blood.2024028005. PMID 40106768